CLINICAL TRIAL: NCT07272551
Title: Investigation of the Effectiveness of the Polyvagal Theory-based Exercise Approach in Chronic Neck Pain
Brief Title: The Effectiveness of the Polyvagal Theory in Chronic Neck Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Mediha Uçan, Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMU-FTR-MU-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Chronic Neck Pain
Keywords: Neck Pain; chronic neck pain; Vagal Nerve Stimulation; Joint Position Sense; Rehabilitation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: The study includes 3 different groups: control, intervention 1 and intervention 2.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Participants in this group will undergo traditional, painless cervical exercises twice a week for 8 weeks. The intervention will not lead to progression, and the same intervention content will be used for 16 sessions. The exercises will be performed by a physical therapist.
  Interventions: Other: Control
- Intervention 1 (Experimental): Participants in this study will undergo exercises based on polyvagal theory twice a week for 8 weeks. The exercise content will be one set. The intervention will not be progressive, and the same intervention content will be used for 16 sessions. The intervention will be administered by a physical therapist.
  Interventions: Other: Intervention 1
- Intervention 2 (Experimental): Participants in this study will receive exercises based on polyvagal theory in addition to traditional, painless cervical exercises twice a week for 8 weeks. Each exercise will be performed for 10 repetitions and 3 sets. Polyvagal theory-based exercises will be performed for 1 set. The intervention will be non-progressive and will use the same intervention content for 16 sessions. The intervention will be administered by a physical therapist.
  Interventions: Other: Intervention 2

INTERVENTIONS:
Other: Control — Participants in this study will undergo traditional, painless cervical exercises twice a week for 8 weeks. Each exercise will be performed for 10 repetitions and 3 sets. The exercises are as follows:
  Traditional, painless cervical exercises will consist of 10 slow repetitions of each of the following cervical movements, starting from a natural resting head position: left rotation, right rotation, flexion, extension, left lateral flexion, and right lateral flexion. Isometric neck exercises will be performed in a straight line forward, backward, right, and left direction, with the patient's own hands providing resistance in the opposite direction.
  Shoulder active ROM exercises will involve participants performing shoulder flexion, abduction up to 90°, and external and internal rotation exercises with their elbows flexed to 90° and their arms at their sides. Additionally, they will be asked to perform shoulder rolls forward and backward while standing.
  Arms: Control
Other: Intervention 1 — In this study, participants will undergo polyvagal theory-based exercises twice a week for 8 weeks, totaling 16 sessions. The exercises are categorized into four main groups: sensory awareness exercises, progressive muscle relaxation, vocalization exercises, and self-soothing touch exercises. Sensory awareness exercises include focused breathing, awareness of upright postures and bodily sensations, lying on the back with eyes closed while focusing on positive thoughts, and walking mindfully in a calm environment. Progressive muscle relaxation involves sequentially tensing and relaxing muscle groups from the toes to the head and visualizing calming scenes through guided imagery. Vocalization exercises consist of tongue trills producing a "ben" sound, humming with a closed mouth, and sustaining vowel sounds. Self-soothing touch exercises include massaging the feet, mindfully touching the arms, face, and palms, and practicing abdominal breathing.
  Arms: Intervention 1
Other: Intervention 2 — Participants in this study will receive exercises based on polyvagal theory in addition to traditional, painless cervical exercises twice a week for 8 weeks. Each exercise will be performed for 3 sets of 10 repetitions. Participants will rest for two seconds after each repetition and five seconds after each set. The exercise content will be the same as described above.
  One set of polyvagal theory-based exercises will be performed. The exercise content will be the same as described above. The intervention will not be progressive, and the same intervention content will be used for 16 sessions. The intervention will be administered by a physiotherapist.
  Arms: Intervention 2

SUMMARY:
This study aimed to examine the effectiveness of a polyvagal theory-based exercise approach on joint position sense, pain, range of motion, functionality, depression, and quality of life in individuals with chronic neck pain.

H0 = The polyvagal theory-based exercise approach has no significant effect on joint position sense, neck pain, range of motion, functionality, depression, or quality of life.

H1 = The polyvagal theory-based exercise approach has a significant effect on joint position sense, neck pain, range of motion, functionality, depression, and quality of life.

DETAILED DESCRIPTION:
Neck pain is one of the most common musculoskeletal problems that negatively impacts individuals' health and quality of life. When chronic painful conditions occur in musculoskeletal disorders, mood disorders such as depression and anxiety can also occur. A long-term history of neck pain is associated with stress, poor quality of life, and decreased functionality.

Polyvagal theory advocates working with the body, becoming aware of it, and connecting with the senses. Exercises based on polyvagal theory can be specifically designed and customized to stimulate the vagus nerve, promote relaxation, and enhance social interaction by following the principles of polyvagal theory.

While polyvagal theory is often used in psychology, it has only been used in rehabilitation in one study, with the potential to improve quality of life by inhibiting the sympathetic nervous system and activating the parasympathetic nervous system, thereby reducing pain perception and stress.

This study, in which participants were divided into three groups: control, intervention 1, and intervention 2, aimed to examine the effectiveness of a polyvagal theory-based exercise approach on joint position sense, pain, range of motion, functionality, depression, and quality of life in individuals with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with chronic neck pain of Grade 1 or 2, lasting at least 3 months
* Individuals whose pain is clinically evaluated and diagnosed
* Individuals with a pain score of 3 or higher on the Visual Analog Scale

Exclusion Criteria:

* Individuals diagnosed with chronic neck pain of Grade 3 or 4
* History of trauma or surgical intervention in the neck region
* Cervical disc herniation, cervical stenosis, or other serious neurological conditions
* Upper extremity radiculopathy
* Acute inflammation or infection
* Severe pathological conditions (e.g., inflammatory diseases, neoplasms, fractures)
* Individuals unable to participate in exercises due to mental or physical impairments
* Pregnancy
* Individuals who have received physiotherapy for chronic neck pain within the last 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Cervical Joint Position Sense | Baseline and after 8 weeks of intervention
  Participants are asked to sit in a chair 90 cm from a white wall. A laser beam is fixed to their head. The laser light on the wall is marked as a reference point. Patients are then asked to turn their heads left and right, one at a time, to the end of the available range, then return to the original position with their eyes open and attempt to align the laser light with the reference point. Their eyes are then closed. As they return their heads to the original position, participants are asked to inform the examiner when they reach the original position. The new laser point on the wall is marked as the target point. Joint position error is calculated in degrees by dividing the arc tangent of the distance between the target and the reference point by 90 cm. The procedure is performed three times for each side for flexion, extension, right-left lateral flexion, and right-left rotation, and the average values of the errors for each side are used for further analysis.

SECONDARY OUTCOMES:
Visual Analog Scale | Baseline and after 8 weeks of intervention
  Neck pain is assessed using a 10-cm Visual Analog Scale. This scale is commonly used in clinical settings to evaluate the effectiveness of pain management. Participants indicate their current pain level by selecting a number between 0 (no pain) and 10 (unbearable pain) along a horizontal line. Previous studies report excellent test-retest reliability.
Joint Range of Motion | Baseline and after 8 weeks of intervention
  Cervical active range of motion is assessed using a standard full-circle goniometer. Measurements are taken with participants seated comfortably in a neutral head position. For flexion and extension, the goniometer axis is placed over the external auditory meatus, the moving arm aligned with the nose, and the stationary arm vertical to the floor. Lateral flexion is measured with the axis on the C7 spinous process, the moving arm aligned with the occipital protuberance and dorsal midline of the head, and the stationary arm along the thoracic spinous processes. For right and left rotation, the axis is placed on the vertex of the head, the stationary arm parallel to a line connecting the acromial processes, and the moving arm directed toward the tip of the nose.
Neck Disability Index (NDI) | Baseline and after 8 weeks of intervention
  Disability is assessed using the Neck Disability Index (NDI) questionnaire. The NDI consists of 10 questions, each with a possible score from 0 to 5. The total score of the 10 questions is divided by the highest possible score, 50, and expressed as a percentage. Higher percentage scores indicate greater disability. The NDI demonstrates good to excellent internal consistency, moderate to excellent reliability, and poor to good responsiveness. The minimum clinically important difference is reported as 20% in a similar cohort of people with chronic neck symptoms.
Beck Depression Inventory (BDI) | Baseline and after 8 weeks of intervention
  his is a 21-item self-report scale that assesses depressive symptoms and attitudes. It provides a four-point Likert-type measurement. It provides information about the severity of depression. Its Turkish adaptation was conducted for reliability and validity by Hisli.
Resting Heart Rate | Immediately before and immediately after each treatment session (for 8 weeks)
  Resting heart rate will be measured after each session using a smartwatch capable of measuring resting heart rate. Measurements will be taken 10 minutes after the exercise session, with patients sitting quietly with an empty bladder. During the measurement, participants will sit with their backs supported and their arms at a 90° angle. Measurements will be made twice, 15 minutes apart, and the average of these two measurements in beats per minute (bpm) will be used.
WHOQOL-BREF | Baseline and after 8 weeks of intervention
  The WHOQOL-BREF is a tool used to assess psychometric properties. It consists of 26 questions related to four domains: physical health, psychological health, social relationships, and environment. Each item is rated on a 5-point Likert scale, with each score ranging from 0 to 100. Interclass correlation coefficients range from 0.71 to 0.91. The WHOQOL BREF is scored for domains. Domain scoring is positive. Higher facet scores indicate higher quality of life. The total raw score is multiplied by 4 to obtain a score comparable to the WHOQOL-100. The total is then converted to a 0-100 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dilanur Kutlu Özkaraoğlu, PhD, Principal Investigator — Istanbul Medipol University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Noi 6:15 studio, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No